CLINICAL TRIAL: NCT03717051
Title: Use of Nicotine Replacement Therapy (NRT) Sample and Brief Smoking Cessation Advice for Recruiting Smokers to Smoking Cessation Services and Motivating Quit Attempts
Brief Title: Use of Nicotine Replacement Therapy (NRT) Sample and Brief Smoking Cessation Advice for Recruiting Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRTsampling2018
Record Dates: First submitted 2018-10-12; First posted 2018-10-23 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation
Keywords: intervention; nicotine replacement sample; smoking cessation; smoking hotspots
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive nicotine replacement therapy (NRT) sampling and medication counseling. The nurse will help the subject to decide which NRT product (patch or gum) he/she can use and advise how to use the NRT based on his/her smoking habit and amount of cigarette consumption. In addition, the nurse will deliver medication counselling which addresses five main components: (1) the benefits for using NRT in quitting, (2) withdrawal symptoms due to smoking cessation, (3) side effects of NRT, (4) instructions for using NRT, and (5) making appointments for TWGHs SC clinics. Afterwards, the participant will receive 1-week free NRT, an education card about NRT and a one-page leaflet provided by the SC clinics.
  Interventions: Drug: Nicotine replacement therapy (NRT) sampling; Behavioral: Medication counseling
- Control (Active Comparator): The control group subjects will receive medication counseling. They will be advised to obtain free NRT by enrolling in the smoking cessation services, but will not be given the sampling. The same one-page leaflet will be provided by the SC clinics.
  Interventions: Behavioral: Medication counseling

INTERVENTIONS:
Drug: Nicotine replacement therapy (NRT) sampling — 1-week free NRT samples (patch or gum)
  Arms: Intervention
Behavioral: Medication counseling — Medication counseling

SUMMARY:
Background More than 60% of the daily smokers in Hong Kong have never tried and have no intention to quit smoking. About 30.8% of daily smokers attempted to quit but failed. Nicotine replacement therapy (NRT) is a safe and effective pharmacotherapy to reduce withdrawal symptoms during early stage of tobacco abstinence and increase quit rate. However, the prevalence of using NRT in Hong Kong is lower than most of the developed countries. The proposed project aims to test if providing free NRT sampling to smokers can increase quit attempt, the use of smoking cessation (SC) services and abstinence.

Methods University undergraduate students will be trained, and will invite smokers at outdoor smoking hotspots to quit smoking and enroll into SC services. Eligible smokers will be randomized to experimental or control group according to a cluster randomization, using recruitment session as the randomization unit. The experimental group will be provided with 1-week free NRT sampling and medication counselling, whereas the control group will be provided medication counselling. Both groups are advised to enroll in the SC services. The primary outcome is the proportion of smokers who report quit attempts at 1 month follow-up

Discussions The findings will inform the feasibility and effectiveness of delivering free NRT sampling to increase quit attempt, the use of smoking cessation services and abstinence. It will yield more information on smokers' adherence to the NRT sampling, side effect and safety issue of the usage.

DETAILED DESCRIPTION:
Study design

The proposed project has 4 phases: (1) Training of SC ambassadors (SCAs) for the SC promotion; (2) SC promotion sessions to deliver the medication counselling and NRT sampling (experimental group), or the advice to use NRT only (control group); (3) Follow-up of the recruited smokers; (4) Evaluation of the effectiveness of training, promotions, and use of NRT sampling. To examine the effectiveness of NRT sampling for recruitment and quitting, a multi-site cluster RCT (allocation ratio 2:1) will be used. All promotion sessions will be randomly allocated to either the experimental or the control group. The experimental group will receive medication counselling and NRT samples, while the control group only receive the advice to use NRT. Both groups are advised to enroll in any smoking cessation service in Hong Kong. Because smokers who receive NRT sampling will be more likely to participate in the study, the experimental sessions will then recruit more smokers than the control sessions. Hence, the allocation ratio of participants is arbitrarily set at 2:1. To increase comparability between the two groups, the promotion sessions of one hotspot will be randomly allocated to either group. All recruitment and quitting outcomes in the smokers between the experimental and control group will be compared.

Subjects

Smokers with the following inclusion criteria will be invited to participate in our RCT: (1) Hong Kong residents, (2) aged 18 to 65 years, (3) have used any tobacco products in the past month, (4) able to read and speak Chinese, (5) have not used NRT for the past month, (6) no severe angina, serious cardiac arrhythmias and hypertension, (7) have not suffered acute myocardial event in the past 4 weeks, (8) neither pregnant nor breastfeeding, (9) not under medication and treatment due to mental illness. To confirm the smoking status, in those who use conventional cigarettes, smokers' exhaled carbon monoxide will be measured on-site. Nurses will measure the blood pressure if smoker is aged over 50 years old, obese by observation, or upon patient requests.

The inclusion criterion no. 3 was "smoke 10 cigarettes or more per day in the past week" and is amended to "have used any tobacco products in the past month". The initial intention of setting the inclusion criteria of at least 10 cigarettes per day (CPD) is to recruit smokers who have moderate to strong level of craving and a greater need for NRT. However, we also recognize that one of the objectives of the research is to promote the use of NRT for quit attempts with NRT sampling. In fact, smokers who smoke less than 10 CPD can also benefit from using NRT gums. Therefore, the change in the inclusion criteria does not deviate from our research aim. In contrast, with the removal of the criterion for CPD, we will be able to reach out to a larger group of smoking population and encourage more smokers to use NRT to quit smoking.

Procedures

In the experimental sessions, the SCAs will approach and distribute souvenirs (e.g. a pen) or leaflets to the smokers at outdoor smoking hotspots for 3-4 hours. The souvenirs and leaflets will have SC messages, quitline number and other SC services. If a smoker is willing to accept them and talk to the SCAs, the SCAs will advise the smoker to quit using the AWARD protocol. The AWARD protocol includes (1) Ask the smoking history, (2) Warn about the high risk (i.e., half of the smokers will die of smoking-related diseases), (3) Advise to quit, (4) Refer to the SC clinics of TWGHs and (5) Repeat the above advice (Do-it-again) [4]. Our previous studies have shown that the AWARD protocol is a feasible and appropriate tool used by non-healthcare professionals to promote smoking cessation [4-6]. If the smoker is interested in smoking cessation, the SCAs will introduce NRT to the smoker and conduct a preliminary assessment of his/her eligibility for enrolling in the "NRT sampling" programme. The SCAs will invite him/her to go to the smoking cessation truck nearby to receive counselling by an onsite nurse. If the smoker is not eligible, he/she can still enroll in the cessation service provided by the SC clinics. The intervention and assessment will mostly be taken place in a smoking cessation truck when the recruitment venues allow us to park the truck nearby, or at outdoor areas when a parking space for a truck is not available.

Intervention: NRT sampling and medication counselling

In the experimental sessions, an onsite nurse will assess whether each participant is fit for using NRT with further assessment on his/her current physical status, medication and blood pressure. If the participant is willing to use NRT to quit smoking and pass the nurse's assessment, he/she will be prescribed the NRT sample, regardless of whether they use NRT for smoking reduction and when the quit day is. The nurse will help the participant decide which type of NRT product (gum: 2mg, patch: 14mg or 21mg) that he/she can use and advise him/her on how to use the NRT based on his/her smoking habit and daily cigarette consumption. In addition, the nurse will deliver medication counselling which addresses five main components: (1) the benefits for using NRT in quitting, (2) withdrawal symptoms due to smoking cessation, (3) side effects of NRT, (4) instructions for using NRT, and (5) making appointments for TWGHs SC clinics. An instruction card for using NRT will be given. Afterwards, the participant will receive 1-week free NRT. Our research staff will send the NRT sample via mail within 2 days.

In the control sessions, all the above procedures for the experimental group will be applied, except that they will not receive an NRT sample and an instruction card about the use of NRT. Instead, they will be advised to obtain free NRT by enrolling in the SC clinics. Both groups will receive a one-page leaflet provided by the SC clinics, and encouraged to make service appointments with the SC clinics. The leaflet briefly introduced this RCT, the use of NRT and the service provided by the smoking cessation clinics.

When the participant has finished the above procedures, the research assistant or trained ambassadors (under supervision of the research staff) or the nurse will introduce the trial of evaluating the effect of NRT sample and the outreach service and screen the eligibility of participating in the trial. If the participant is eligible, the research assistant will seek his/her consent to participate in the trial, and complete a baseline questionnaire.

Some smokers are willing to participate in the RCT, but they have no time to receive all intervention or complete all recruitment procedures at the hotspots. In these cases, the SCAs will only briefly introduce the RCT, ask the participants to give written consent. A nurse will contact these participants to complete the baseline questionnaire and deliver the intervention (medication advice and NRT prescription) within the same day. If the participants are in the experimental group, after the telephone counselling by the nurse, our research staff will send the NRT sample via mail within 2 days.

Randomization

We will use cluster randomization based on promotion session as the cluster unit because the procedures of individual randomization are difficult in outdoor areas as found in our pilot RCT. The PI will randomly allocate the promotion sessions within a hotspot to the 2 groups by a list of group allocation which is based on a list of random numbers from Excel programme. Each hotspot will have 2 or more promotion sessions, and each session will last for about 3-4 hours. If a hotspot has 2 promotion sessions on 1 single day, the 2 sessions will be allocated into the same RCT group, and we will organize 2 more promotion sessions in this hotspot on another day.

Allocation concealment

All recruitment staff will know the group allocation before each promotion session, so no group concealment can be done.

Blinding

Participants, recruitment staff and nurses cannot and will not be blinded to the intervention. Assessors of the follow-up outcomes and the research analysts will not be involved in the recruitment and intervention delivery, and will be blinded to the group allocation (single blindness).

Baseline assessments

Baseline information includes socio-demographics, current use of conventional and new tobacco products, such as heat-not-burn tobacco products and electronic cigarettes, history of quit attempts, and intention to quit. Nicotine dependence will be assessed by the Fagerström Test for Nicotine Dependence.24 Participants will also be asked about their self-efficacy in quitting, based on the perceived importance, difficulty and confidence to quit smoking on a Likert scale from 0 to 10.

Follow-up

All the smokers who consent to the follow-up will be contacted via telephone or WhatsApp around one week by a nurse or a trained research staff after recruitment. The aim of this follow-up is (1) to enquire if there is any progress towards smoking cessation and (2) encourage the use of NRT for a quit attempt and/or enrollment in SC services as soon as possible. If participants show no interest to quit, the nurse/research staff will use the "5R" approach to re-motivate the quitting intention. The "5R" approach is being adopted by the local and international smoking cessation guideline including the discussion on why quitting is important (relevance), hazards of smoking (risk), benefits of quitting (rewards), difficulties (roadblocks) and repeated quit attempts (repetition). If participants report any contra-indication(s) to NRT, the nurse/research staff will discuss the reasons with them, and, if necessary, refer the participants to the physician in the smoking cessation clinic.

At 1-, 3- and 6-month follow-up, the quitting outcomes will be assessed by a trained interviewer through telephone who is blinded to the subject's group status. A small amount (HK$50=US$6.4) of cash voucher will be offered to those who completed a follow-up survey. At 6-month follow-up, participants who reported no smoking in past 7 days will be invited for a biochemical validation of the abstinence. Participants with exhaled carbon monoxide 4ppm or below and saliva cotinine level below 10ng/ml will be considered as validated abstinence. Participants of the biochemical validation, no matter the abstinence status is confirmed, will be offered a HK$50 (US$6.4) cash voucher for the travel compensation.

Sample size determination

As we predicted that the recruitment sessions of providing free NRT samples will recruit more smokers, participant ratio of the 2 trial groups is arbitrarily set at 2:1. At the time we designed this trial, our preliminary analysis of the aforementioned pilot RCT showed that the rate of quit attempt in the intervention and control group was 26% and 12% at 3-month follow-up, respectively. We arbitrarily reduced these rates to 20% and 8% for 1-month follow-up. To detect a significant difference with normal test and a power of 95% and 5% significance level, we need 485 subjects in the RCT (allocation ratio 2:1; 323 vs 162). Based on the method of Eldridge et al. (2006),29 conservatively assuming that we could recruit 8 participants per session on average and the intra-cluster correlation coefficient was 0.1, the design effect is estimated to be 1.7. Thus, the minimum sample size required for the trial is 825 (=1.7 X 485) participants and 104 sessions in total. With the similar calculation, the required sample size for detecting a significant difference in the proportion of using any smoking cessation service is 421.

Statistical analysis

An independent data analyst will perform the data check of missing, duplication and validity on the completed dataset before analysis is done. All data will be de-identified in the data analysis. To assess the effect of NRT sampling to the process outcomes, the number of smokers who accept the brief advice or consent the RCT in each recruitment session will be the outcome variables of Poisson regression model, with group allocation as the predictor, and total number of approached smokers in that promotion session as the offset variable. Considering the possibility of correlated outcomes of participants within the recruitment session, an analysis by generalized estimating equations model, assigning session as a random effect, will be used to summarize the intervention effect on the primary outcome. The analysis adopted a longitudinal approach with an exchangeable structure for the correlation matrix of the outcome. Other secondary outcomes will be analyzed with either generalized estimating equations models (binary outcomes; e.g. tobacco abstinence) or linear mixed model (continuous outcomes; e.g. perceived importance to quit smoking). Both intention-to-treat (treating participants as smokers without quit attempts and no use of cessation services if they are lost to follow-up) and per protocol analysis will be done. Subgroup analysis of comparing the primary and secondary outcomes between participants receiving the nurse-led intervention onsite and those receiving the intervention via telephone will be done.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* aged 18 to 65 years
* have used any tobacco products in the past month
* able to read and speak Chinese
* have not used NRT for the past month

Exclusion Criteria:

* Have severe angina, serious cardiac arrhythmias and hypertension
* Have suffered from acute myocardial event in the past 4 weeks
* Pregnant nor breastfeeding
* Under medication and treatment due to mental illness

One of the inclusion criteria was "smoke 10 cigarettes or more per day in the past week" and is amended to "have used any tobacco products in the past month". The initial intention of setting the inclusion criteria of at least 10 cigarettes per day (CPD) is to recruit smokers who have moderate to strong level of craving and a greater need for NRT. However, we also recognize that one of the objectives of the research is to promote the use of NRT for quit attempts with NRT sampling. In fact, smokers who smoke less than 10 CPD can also benefit from using NRT gums. Therefore, the change in the inclusion criteria does not deviate from our research aim. In contrast, with the removal of the criterion for CPD, we will be able to reach out to a larger group of smoking population and encourage more smokers to use NRT to quit smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2018-10-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Derek Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Background] Cropsey KL, Trent LR, Clark CB, Stevens EN, Lahti AC, Hendricks PS. How low should you go? Determining the optimal cutoff for exhaled carbon monoxide to confirm smoking abstinence when using cotinine as reference. Nicotine Tob Res. 2014 Oct;16(10):1348-55. doi: 10.1093/ntr/ntu085. Epub 2014 Jun 2. PMID 24891552
- [Background] Montalto NJ, Wells WO. Validation of self-reported smoking status using saliva cotinine: a rapid semiquantitative dipstick method. Cancer Epidemiol Biomarkers Prev. 2007 Sep;16(9):1858-62. doi: 10.1158/1055-9965.EPI-07-0189. PMID 17855706
- [Background] Chan SSC, Cheung YTD, Wong YMB, Kwong A, Lai V, Lam TH. A Brief Smoking Cessation Advice by Youth Counselors for the Smokers in the Hong Kong Quit to Win Contest 2010: a Cluster Randomized Controlled Trial. Prev Sci. 2018 Feb;19(2):209-219. doi: 10.1007/s11121-017-0823-z. PMID 28755244
- [Background] Chan SS, Wong DC, Cheung YT, Leung DY, Lau L, Lai V, Lam TH. A block randomized controlled trial of a brief smoking cessation counselling and advice through short message service on participants who joined the Quit to Win Contest in Hong Kong. Health Educ Res. 2015 Aug;30(4):609-21. doi: 10.1093/her/cyv023. Epub 2015 Jun 25. PMID 26116584
- [Background] Cheung YTD, Lam TH, Li WHC, Wang MP, Chan SSC. Feasibility, Efficacy, and Cost Analysis of Promoting Smoking Cessation at Outdoor Smoking "Hotspots": A Pre-Post Study. Nicotine Tob Res. 2018 Nov 15;20(12):1519-1524. doi: 10.1093/ntr/ntx147. PMID 28655173
- [Background] Cheung YT, Wang MP, Li HC, Kwong A, Lai V, Chan SS, Lam TH. Effectiveness of a small cash incentive on abstinence and use of cessation aids for adult smokers: A randomized controlled trial. Addict Behav. 2017 Mar;66:17-25. doi: 10.1016/j.addbeh.2016.11.006. Epub 2016 Nov 10. PMID 27863323
- [Background] Abdullah AS, Hedley AJ, Chan SS, Lam TH. A randomized controlled trial of two different lengths of nicotine replacement therapy for smoking cessation. Biomed Res Int. 2013;2013:961751. doi: 10.1155/2013/961751. Epub 2013 Sep 9. PMID 24089693
- [Background] Census & Statistics Department (Hong Kong SAR government). Thematic Household Survey, Report No. 59: Pattern of Smoking. Hong Kong: Census & Statistics Department 2016.
- [Background] Lam TH. Absolute risk of tobacco deaths: one in two smokers will be killed by smoking: comment on "Smoking and all-cause mortality in older people". Arch Intern Med. 2012 Jun 11;172(11):845-6. doi: 10.1001/archinternmed.2012.1927. No abstract available. PMID 22688993
- [Background] Leung DYP, Chan SSC, Jiang CQ, et al. Providing Smoking Cessation Services and Its Relationship with Knowledge and Attitudes: A Comparison of the Guangzhou and Hong Kong Nurses. Journal of Comparative Asian Development 2009;8(1):179-205.
- [Background] Lam TH, Jiang C, Chan YF, Chan SS. Smoking cessation intervention practices in Chinese physicians: do gender and smoking status matter? Health Soc Care Community. 2011 Mar;19(2):126-37. doi: 10.1111/j.1365-2524.2010.00952.x. Epub 2010 Sep 9. PMID 21309876
- [Background] Aveyard P, Foulds J. The 2009 US Clinical Practice Guideline: the key recommendations and a commentary (www.treatobacco.net 2009 Ask the Experts). 2009 Date;Volume. http://www.treatobacco.net/fr/page_349.php (accessed 01 March 2009).
- [Background] Leung DY, Chan SS, Chan V, Lam TH. Hardcore smoking after comprehensive smoke-free legislation and health warnings on cigarette packets in Hong Kong. Public Health. 2016 Mar;132:50-6. doi: 10.1016/j.puhe.2015.10.007. Epub 2015 Nov 21. PMID 26612457
- [Background] Chan SSC, Cheung YTD, Wan Z, Wang MP, Lam TH. Proactive and Brief Smoking Cessation Intervention for Smokers at Outdoor Smoking "Hotspots" in Hong Kong. J Cancer Educ. 2018 Apr;33(2):365-370. doi: 10.1007/s13187-016-1085-3. PMID 27474113
- [Background] Kasza KA, Hyland AJ, Borland R, McNeill AD, Bansal-Travers M, Fix BV, Hammond D, Fong GT, Cummings KM. Effectiveness of stop-smoking medications: findings from the International Tobacco Control (ITC) Four Country Survey. Addiction. 2013 Jan;108(1):193-202. doi: 10.1111/j.1360-0443.2012.04009.x. Epub 2012 Aug 14. PMID 22891869
- [Background] West R, Raw M, McNeill A, Stead L, Aveyard P, Bitton J, Stapleton J, McRobbie H, Pokhrel S, Lester-George A, Borland R. Health-care interventions to promote and assist tobacco cessation: a review of efficacy, effectiveness and affordability for use in national guideline development. Addiction. 2015 Sep;110(9):1388-403. doi: 10.1111/add.12998. PMID 26031929
- [Background] Borland R, Li L, Driezen P, Wilson N, Hammond D, Thompson ME, Fong GT, Mons U, Willemsen MC, McNeill A, Thrasher JF, Cummings KM. Cessation assistance reported by smokers in 15 countries participating in the International Tobacco Control (ITC) policy evaluation surveys. Addiction. 2012 Jan;107(1):197-205. doi: 10.1111/j.1360-0443.2011.03636.x. PMID 21883605
- [Background] Beard E, Brown J, Michie S, Kaner E, Meier P, West R. Use of aids for smoking cessation and alcohol reduction: A population survey of adults in England. BMC Public Health. 2016 Dec 8;16(1):1237. doi: 10.1186/s12889-016-3862-7. PMID 27931202
- [Background] Barnoya J, Jin L, Hudmon KS, Schootman M. Nicotine replacement therapy, tobacco products, and electronic cigarettes in pharmacies in St. Louis, Missouri. J Am Pharm Assoc (2003). 2015 Jul-Aug;55(4):405-12. doi: 10.1331/JAPhA.2015.14230. PMID 26115460
- [Background] Carpenter MJ, Hughes JR, Gray KM, Wahlquist AE, Saladin ME, Alberg AJ. Nicotine therapy sampling to induce quit attempts among smokers unmotivated to quit: a randomized clinical trial. Arch Intern Med. 2011 Nov 28;171(21):1901-7. doi: 10.1001/archinternmed.2011.492. PMID 22123796
- [Background] Jardin BF, Cropsey KL, Wahlquist AE, Gray KM, Silvestri GA, Cummings KM, Carpenter MJ. Evaluating the effect of access to free medication to quit smoking: a clinical trial testing the role of motivation. Nicotine Tob Res. 2014 Jul;16(7):992-9. doi: 10.1093/ntr/ntu025. Epub 2014 Mar 7. PMID 24610399
- [Background] Cunningham JA, Kushnir V, Selby P, Tyndale RF, Zawertailo L, Leatherdale ST. Effect of Mailing Nicotine Patches on Tobacco Cessation Among Adult Smokers: A Randomized Clinical Trial. JAMA Intern Med. 2016 Feb;176(2):184-90. doi: 10.1001/jamainternmed.2015.7792. PMID 26809849
- [Background] Cheung YT, Leung JP, Cheung CK, Li WH, Wang MP, Lam TH. Motivating smokers at outdoor public smoking hotspots to have a quit attempt with a nicotine replacement therapy sample: study protocol for a randomized controlled trial. Trials. 2016 Jul 26;17(1):355. doi: 10.1186/s13063-016-1485-z. PMID 27456342
- [Background] Eldridge SM, Ashby D, Kerry S. Sample size for cluster randomized trials: effect of coefficient of variation of cluster size and analysis method. Int J Epidemiol. 2006 Oct;35(5):1292-300. doi: 10.1093/ije/dyl129. Epub 2006 Aug 30. PMID 16943232
- [Background] Flocke SA, Step MM, Lawson PJ, Smith S, Zyzanski SJ. Development of a Measure of Incremental Behavior Change Toward Smoking Cessation. Nicotine Tob Res. 2017 Dec 13;20(1):73-80. doi: 10.1093/ntr/ntw217. PMID 27613910
- [Background] Wang MP, Suen YN, Li WH, Lam CO, Wu SY, Kwong AC, Lai VW, Chan SS, Lam TH. Intervention With Brief Cessation Advice Plus Active Referral for Proactively Recruited Community Smokers: A Pragmatic Cluster Randomized Clinical Trial. JAMA Intern Med. 2017 Dec 1;177(12):1790-1797. doi: 10.1001/jamainternmed.2017.5793. PMID 29059277
- [Derived] Cheung YTD, Chan CHH, Ho KS, Tang C, Lau CWH, Li WHC, Wang MP, Lam TH. Effectiveness of nicotine replacement therapy sample at outdoor smoking hotspots for initiating quit attempts and use of smoking cessation services: a protocol for a cluster randomised controlled trial. BMJ Open. 2020 Apr 7;10(4):e036339. doi: 10.1136/bmjopen-2019-036339. PMID 32269028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started from July 1st, 2018 to June 30th, 2020. Participants of this study were recruited at outdoor smoking hotspots in Hong Kong.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 352 | 482
Completed | 352 | 482
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 482 | 352 | 834
Age, Continuous [Mean (Full Range); unit: years] | 40.54 [18 to 74] | 41.33 [18 to 65] | 40.87 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 57 | 156
  Male | 383 | 295 | 678
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 482 | 352 | 834
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Enroll in Any Smoking Cessation Service in Hong Kong
Description: Number of participants who enroll in any smoking cessation service in Hong Kong
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 156 | 158

2. Primary Outcome: Number of Participants With Self-reported Quit Attempt
Description: No smoking for at least 24 hours in the past month
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 214 | 153

3. Secondary Outcome: Number of Participants Who Enroll in Any Smoking Cessation Service in Hong Kong
Description: Number of participants who enroll in any smoking cessation service in Hong Kong
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 247 | 213

4. Secondary Outcome: Number of Participants With Self-reported Quit Attempt
Description: No smoking for at least 24 hours in the past month
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 300 | 243

5. Secondary Outcome: Number of Participants With Self-reported Use of NRT in Past Week/Month
Description: self-reported use of NRT in past week/month
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 192 | 121

6. Secondary Outcome: Number of Participants With Self-reported Use of NRT in Past Week/Month
Description: self-reported use of NRT in past week/month
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 92 | 86

7. Secondary Outcome: Number of Participants With Self-reported Tobacco Abstinence in Past 7 Days
Description: self-reported tobacco abstinence in past 7 days
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 95 | 79

8. Secondary Outcome: Number of Participants With Self-reported Tobacco Abstinence in Past 30 Days
Description: self-reported tobacco abstinence in past 30 days
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 68 | 52

9. Secondary Outcome: Number of Participants With Self-reported Tobacco Abstinence in Past 7 Days
Description: self-reported tobacco abstinence in past 7 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 104 | 92

10. Secondary Outcome: Number of Participants With Self-reported Tobacco Abstinence in Past 30 Days
Description: self-reported tobacco abstinence in past 30 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 93 | 77

11. Secondary Outcome: Biochemically Validated Abstinence at 6-month Follow-up
Description: measurement of exhaled carbon monoxide using a Smokerlyzer, and a saliva cotinine test
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
Participants | 22 | 10

12. Secondary Outcome: Perceived Importance, Difficulty and Confidence to Quit Smoking
Description: Self-efficacy will be evaluated according to the importance of quitting on a scale of 0 to 10 (0, least important; 10, most important), the difficulty of quitting on a scale of 0 to 10 (0, least difficult; 10, most difficult), and confidence in quitting on a scale of 0 to 10 (0, least confident; 10, most confident). For the scale of measuring quitting importance and confidence, higher scores mean a better outcome and for the scale of measuring difficulty, higher scores mean a worse outcome.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
score on a scale
  Importance | 7.60 (2.30) | 7.88 (2.09)
  Difficulty | 7.02 (2.42) | 7.38 (2.33)
  Confidence | 6.39 (2.66) | 6.97 (2.43)

13. Secondary Outcome: Perceived Importance, Difficulty and Confidence to Quit Smoking
Description: Self-efficacy will be evaluated according to the importance of quitting on a scale of 0 to 10 (0, least important; 10, most important), difficulty of quitting on a scale of 0 to 10 (0, least difficult; 10, most difficult), and confidence in quitting on a scale of 0 to 10 (0, least confident; 10, most confident)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
score on a scale
  Importance | 7.80 (2.15) | 7.53 (2.26)
  Difficulty | 7.25 (2.38) | 7.34 (2.18)
  Confidence | 6.58 (2.50) | 6.47 (2.49)

14. Secondary Outcome: Perceived Importance, Difficulty and Confidence to Quit Smoking
Description: as for outcome 13
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
score on a scale
  Importance | 7.36 (2.46) | 8.09 (2.02)
  Difficulty | 7.53 (2.19) | 7.22 (2.46)
  Confidence | 6.02 (2.87) | 6.47 (2.95)

15. Secondary Outcome: Progression Towards Smoking Cessation
Description: progression towards smoking cessation as measured by Incremental Behavior Change toward Smoking cessation (IBC-S). The minimum value is 3 and the maximum value is 27. Higher scores mean a better outcome.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
score on a scale | 16.04 (3.24) | 15.12 (3.30)

16. Secondary Outcome: Progression Towards Smoking Cessation
Description: as for outcome 15
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
score on a scale | 14.60 (2.99) | 14.42 (3.00)

17. Secondary Outcome: Progression Towards Smoking Cessation
Description: as for outcome 15
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 482 | 352
score on a scale | 13.94 (2.85) | 14.58 (2.77)

ADVERSE EVENTS:
Time Frame: 6 months
Description: For the benefit of our research staff and participants, we will report all adverse events.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/482 | 0/352
Serious Adverse Events (participants affected / at risk) | 0/482 | 0/352
Other Adverse Events (participants affected / at risk) | 0/482 | 0/352

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03717051/Prot_SAP_000.pdf